CLINICAL TRIAL: NCT00825019
Title: A Double-Blind, Multicenter Study Evaluating the Efficacy and Safety of One Fixed Dose of SR58611A (700 mg/Day) Versus Placebo and Paroxetine (20 mg/Day) in Patients With a Recurrent Major Depressive Episode.
Brief Title: Efficacy and Safety of One Single Dose of SR58611 Compared to Placebo and Paroxetine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5379
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorders
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — amibegron; Amibegron hydrochloride; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: amibegron (SR58611A)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo
- 3 (Active Comparator): paroxetine
  Interventions: Drug: paroxetine

INTERVENTIONS:
Drug: amibegron (SR58611A) — oral administration of 2x 700 mg/day in 12h intervals
  Arms: 1
Drug: placebo — oral administration in 12h intervals
  Arms: 2
Drug: paroxetine — oral administration of 20 mg/day
  Arms: 3

SUMMARY:
Primary objective is to demonstrate the antidepressant efficacy on the Hamilton depression rating scale (HAM-D) of amibegron (SR58611) 700 mg/day compared to placebo in the treatment of patients with a recurrent major depressive episode (MDD).

Secondary objective is to assess the safety profile of amibegron 700 mg/d in comparison to placebo and to assess plasma concentrations of the active metabolite.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from a recurrent major depressive episode of at least moderate intensity (DSM-IV)
* patients have been hospitalized for the treatment of a previous episode, or a previous episode required antidepressant treatment(s)at the recommended dose level for at least 2 months.
* the duration of the current episode is of at least six weeks unless the severity of symptoms justifies shorter duration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2003-09; Primary Completion 2004-10 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
change from baseline of the total score of the HAM-D 17 items | 6 weeks

SECONDARY OUTCOMES:
HAM-D subscores, HAMD responders and remitters, HAM-A total score and subscores | 6 weeks
Montgomery-Asberg Depression Rating Scale (MADRS) total score | 6 weeks
clinical global impression (CGI) severity and improvement scores | 6 weeks
patient global impression (PGI) improvement score | 6 weeks
social and occupational functioning assessment scale (SOFAS) score | 6 weeks
AEs, Arizona Sexual Experience Scale (ASEX), | 6 weeks
laboratory parameters, physical examination findings, ECG parameters, change of vital signs, body weight | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States